CLINICAL TRIAL: NCT00275912
Title: A 24-week Prospective Open-label Multicenter Study to Evaluate the Effect on Seizure Frequency, Safety and Tolerability of Oxcarbazepine Monotherapy in Children With Partial Seizures
Brief Title: Efficacy, Safety, and Tolerability of Oxcarbazepine Monotherapy in Children With Partial Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRI476BRU02
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Epilepsy, Partial Seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oxcarbazepine

SUMMARY:
This study is aimed to collect additional data regarding the efficacy in reducing the frequency of partial seizures, as well as the safety and tolerability, of oxcarbazepine monotherapy in children.

ELIGIBILITY:
Inclusion Criteria:

* males and females, 6 months - 17 years of age;
* diagnosis of epilepsy, partial seizures;
* ineffective or intolerable present therapy with 1 antiepileptic drug, or none of previous antiepileptic therapy

Exclusion Criteria:

* progressive lesion of brain revealed by CT/MRI that performed no earlier than 2 years prior to screening;
* non-epileptic seizures;
* drug or alcohol dependence during a year prior to screening;

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 6 Months to 17 Years | Sex: All
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2006-09-11 (Actual); Primary Completion 2007-09-28 (Actual); Study Completion 2007-09-28 (Actual)

PRIMARY OUTCOMES:
Epileptic activity at electroencephalography in rest
Flash light and hyperventilation test with electroencephalography
Frequency of epileptic episodes according to patient's diary
Electrocardiogram analysis for rhythm and conduction
Blood test for sodium, hepatic enzymes and blood cells

SECONDARY OUTCOMES:
Tolerability and safety of 24 week's treatment with oxcarbazepine monotherapy in children with partial seizures
Rate of patients with total and partial control of epilepsy
Rate of patients requiring additional antiepileptic drugs

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (5):
- Russia (5):
  - Moscow Scientific Research Institute of Pediatrics and Pediatric Surgery, Moscow
  - Russian State Medical University clinically based on Russian Pediatric Clinical Hospital, Moscow
  - Scientific-practical centre of children treatment suffering from craniofacial malformation and congenital pathology of nervous system, Moscow
  - St. Petersburg State Pediatrics Medical Academy, Saint Petersburg
  - Regional Pediatric Clinical Hospital №1 EkaterinburgRegional Pediatric Clinical Hospital №1, Yekaterinburg